CLINICAL TRIAL: NCT06374394
Title: A Phase 3, Open-label, Randomized, Controlled Study to Evaluate the Immune Response, Safety and Reactogenicity of RSVPreF3 OA Investigational Vaccine When Co-Administered With a COVID-19 mRNA Vaccine (Omicron XBB.1.5) in Adults Aged 50 Years and Above
Brief Title: A Study on the Immune Response and Safety of a Vaccine Against Respiratory Syncytial Virus (RSV) When Given Alone and Together With a COVID-19 mRNA Vaccine in Adults Aged 50 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217848; 2023-510196-59-00 (Other: EU CTR Number)
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; Respiratory Syncytial Virus; COVID-19 mRNA vaccine; Immunogenicity; Safety; Reactogenicity; Older Adults
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Co-Ad Group (Experimental): Participants received a single dose of RSVPreF3 OA vaccine and a single dose of COVID-19 mRNA vaccine at Day 1, in different arms.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: COVID-19 mRNA vaccine
- Control Group (Active Comparator): Participants received a single dose of COVID-19 mRNA vaccine at Day 1, followed by a single dose of RSVPreF3 OA vaccine at Day 31.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: COVID-19 mRNA vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — 1 dose of RSVPreF3 OA investigational vaccine is administered intramuscularly on Day 1 to participants in the Co-ad Group and on Day 31 to participants in the Control Group.
Biological: COVID-19 mRNA vaccine — 1 dose of COVID-19 mRNA vaccine is administered intramuscularly on Day 1 to participants in the Co-ad and Control Groups.

SUMMARY:
This study is assessing the immunogenicity, safety and reactogenicity of the RSVPreF3 OA investigational vaccine when it is co-administered with a COVID-19 messenger ribonucleic acid (mRNA) vaccine (Omicron XBB.1.5), compared to administration of the vaccines separately in adults aged 50 years and above.

ELIGIBILITY:
Inclusion Criteria:

• Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).

Note: In case of physical incapacity that would preclude the self-completion of the diary cards, either site staff can assist the participant (for activities performed during site visits) or the participant may assign a caregiver to assist him/her with this activity (for activities performed at home). However, at no time will the site staff or caregiver evaluate the participant's health status while answering diaries or make decisions on behalf of the participant.

* Written or witnessed informed consent obtained from the participant (participant must be able to understand the informed consent) prior to performance of any study-specific procedure.
* A male/female of ≥50 Years of age (YOA) at the time of the first study intervention administration.
* Participants who are medically stable in the opinion of the investigator at the time of first vaccination. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.

A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.

• Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.

Participants who have received previously a SARS-CoV-2 vaccine, being administered at least 3 months prior to study vaccination.

* Female participants of non-childbearing potential may be enrolled in the study. Non childbearing potential is defined as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, and post-menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant.

  * has practiced adequate contraception from 1 month prior to study intervention administration and agreed to continue adequate contraception for at least 1 month after the last vaccination.
  * has a negative pregnancy test on the day of and prior to study intervention administration.

Exclusion Criteria:

Medical Conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions, including a known history of severe allergic reaction (e.g., anaphylaxis).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, resulting from disease (e.g., current malignancy, human immunodeficiency virus) or immunosuppressive/cytotoxic therapy (e.g., medication used during cancer chemotherapy, organ transplantation, or to treat autoimmune disorders), based on medical history and physical examination (no laboratory testing required).
* Any history of myocarditis or pericarditis.
* Recurrent history or uncontrolled neurological disorders or seizures. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol (e.g. completion of diary cards, attend regular phone calls/study site visits).
* Serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival up to study end).
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any SAE attributed to a previous dose of the SARS-CoV-2 mRNA vaccine.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Recent SARS-CoV-2 infection within 3 months prior to the COVID-19 vaccine dose administration. Timelines to be determined from symptoms onset or positive COVID-19 test (if infection was asymptomatic).

Prior/Concomitant Therapy Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study interventions during the period beginning 30 days before the first dose of study interventions and ending 30 days after the last vaccine administration, or their planned use during the study period.

* Planned administration of a vaccine in the period starting 30 days before the first dose and ending 30 days after the last dose of study intervention(s) administration*, with the exception of inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after the study vaccination.

  *If emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine, provided it is used according to the local governmental recommendations and Sponsor is notified.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the last blood sampling visit.

  * Up to 3 months prior to the study intervention administration:

    * For corticosteroids, this will mean prednisone equivalent ≥ 20 mg/day. Inhaled and topical steroids are allowed.
    * Administration of immunoglobulins and/or any blood products or plasma derivatives.
  * Up to 6 months prior to study intervention administration: long-acting immune modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies and antitumoral medication.
* Administration of any SARS-CoV-2 vaccine during the 3 months preceding the study COVID-19 mRNA vaccine administration.
* Previous vaccination with licensed or investigational RSV vaccine. Prior/Concurrent Clinical Study Experience
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other Exclusion Criteria

* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Participation of any study personnel or their immediate dependents, family, or household members.
* Planned move during the study conduct that prohibits participation until study end.
* Bedridden participants.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (8):
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Newport News, Virginia
- Belgium (5):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kluisbergen
  - GSK Investigational Site, Mechelen
- Netherlands (4):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zutphen
- Spain (4):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Boadilla Del Monte Madrid
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 841 enrolled participants, 833 participants were randomized in a 1:1 ratio to either Co-Ad Group or Control Group at Day 1 and started the study. These participants were included in the Exposed Set.
Period: Overall Study
Arm/Group | Co-Ad Group | Control Group
Started | 417 | 416
Completed | 409 | 398
Not Completed | 8 | 18
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 6 | 9
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Exposed set included all participants that received at least one study administration dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Ad Group | Control Group | Total
Number analyzed (Participants) | 417 | 416 | 833
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 63.7 (8.4) | 63.5 (8.4) | 63.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 223 | 439
  Male | 201 | 193 | 394
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — American Indian or Alaska Native and Asian are considered as minority races in this study and are presented together as "Other Races".
  Participants
    Other Races | 5 | 7 | 12
    White | 378 | 375 | 753
    Black or African American | 31 | 32 | 63
    Multiple | 1 | 1 | 2
    Not reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean Titers (GMT) of Respiratory Syncytial Virus-A (RSV-A) Neutralizing Titers at 1 Month After the RSVPreF3 OA Vaccination
Description: RSV-A neutralizing titers were provided as group GMTs and expressed as estimated dilution 60 (ED60) titers. Adjusted GMTs are derived using an ANCOVA model on log10-transformed titers for the neutralization assay. The final ANCOVA model adjusted for baseline differences (in the pre-dose titers) includes treatment group and age category (age at vaccination: 50-59, 60-69 or ≥70 years) as fixed effects, and the pre-dose log10-transformed titers as a covariate.
Time Frame: At 1 month post-RSVPreF3 OA vaccine dose administration (at Day 31 for Co-Ad Group and Day 61 for Control Group)
Population: Per protocol set (PPS) for RSVPreF3 OA included participants who: received RSVPreF3 OA, had immunogenicity results for RSV titers, complied with the blood draw interval, without intercurrent medical conditions, without prohibited concomitant medication/vaccination, did not meet criteria for elimination. Only participants included in both pre-vaccination and 1-month post vaccination timepoints and with results for adjusted GMTs for RSV-A at 1-month post dose were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 382 | 364
Titers | 7885.8 [7168.1 to 8675.3] | 8803.4 [7985.0 to 9705.7]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate non-inferiority of humoral immune response to RSVPreF3 OA vaccine when co-administered with a COVID-19 mRNA vaccine compared to RSVPreF3 OA vaccine administered alone; Test type: Non-Inferiority — Non-inferiority (NI) was to be demonstrated if the upper limit of the 2-sided 95% confidence interval (CI) of the GMT ratio between the Control Group (at Day 61) versus Co-Ad Group (at Day 31) for RSV-A neutralizing titers 1-month after the RSVPreF3 OA vaccine dose was less than or equal to (≤) 1.5; ANCOVA; ANCOVA model included the treatment group and age category at vaccination as fixed effects and the pre-dose log10 titer as covariate; Geometric Mean Ratio (GMR) = 1.12, 95% CI 2-sided [0.97 to 1.28] — The GMR is based on the back transformation of the group comparisons in the ANCOVA model applied to the logarithmically-transformed titers

2. Primary Outcome: Adjusted GMTs of RSV-B Neutralizing Titers at 1 Month After the RSVPreF3 OA Vaccination
Description: RSV-B neutralizing titers were provided as group GMTs and expressed as estimated dilution 60 (ED60) titers. Adjusted GMTs are derived using an ANCOVA model on log10-transformed titers for the neutralization assay. The final ANCOVA model adjusted for baseline differences (in the pre-dose titers) includes treatment group and age category (age at vaccination: 50-59, 60-69 or ≥70 years) as fixed effects, and the pre-dose log10-transformed titers as a covariate.
Time Frame: At 1 month post-RSVPreF3 OA vaccine dose administration (at Day 31 for Co-Ad Group and Day 61 for Control Group)
Population: Analysis was performed on PPS for RSVPreF3 OA. Only participants included in both pre-vaccination and 1-month post vaccination timepoints and with results for adjusted GMTs for RSV-B at 1-month post dose were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 382 | 364
Titers | 7333.3 [6678.6 to 8052.0] | 7903.1 [7182.6 to 8695.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2-sided 95% CI of the GMT ratio between the Control Group (at Day 61) versus Co-Ad Group (at Day 31) for RSV-B neutralizing titers 1-month after the RSVPreF3 OA vaccine dose was ≤1.5; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMR = 1.08, 95% CI 2-sided [0.94 to 1.23] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Adjusted GMTs of SARS-CoV-2 Omicron XBB.1.5 Neutralizing Titers at 1 Month After the COVID-19 mRNA Vaccination
Description: SARS-CoV-2 Omicron XBB.1.5 neutralizing titers against the pseudovirus bearing S protein were provided as group GMTs and expressed as titers. The neutralizing titer was calculated as the reciprocal serum dilution corresponding to the 50% signal reduction (NT50). Adjusted GMTs are derived using an ANCOVA model on log10-transformed titers for the neutralization assay. The final ANCOVA model adjusted for baseline differences (in the pre-dose titers) includes treatment group and age category (age at vaccination: 50-59, 60-69 or ≥70 years) as fixed effects, and the pre-dose log10-transformed titers as a covariate.
Time Frame: At 1 month post-COVID-19 mRNA vaccine dose administration (at Day 31 for both groups)
Population: The PPS for COVID-19 mRNA included participants who:received COVID-19 mRNA, had immunogenicity results for SARS-CoV-2 titers, complied with the blood draw interval, without intercurrent medical conditions, without prohibited concomitant medication/vaccination, did not meet criteria for elimination. Only participants included in both pre-vaccination and 1-month post vaccination timepoints and with results for adjusted GMTs for SARS-CoV-2 titers at 1-month post dose were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 380 | 381
Titers | 1063.6 [960.2 to 1178.2] | 1392.0 [1256.9 to 1541.5]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate non-inferiority of humoral immune response to a COVID-19 mRNA vaccine when co-administered with the RSVPreF3 OA vaccine compared to COVID-19 mRNA vaccine administered alone; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2-sided 95% CI of the GMT ratio between the Control Group (at Day 31) versus Co-Ad group (at Day 31) for SARS-CoV-2 neutralizing titers 1-month after the COVID-19 mRNA vaccine dose was ≤1.5; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMR = 1.31, 95% CI 2-sided [1.13 to 1.51] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: RSV-A Neutralizing Titers Expressed as GMT at 1 Month After RSVPreF3 OA Vaccination
Description: Neutralizing titers for RSV-A were measured with neutralizing assay and the results were expressed as GMT. GMT is a descriptive statistic calculated directly from the observed titer values at the 1-month post-vaccination timepoint for all participants in the analysis set, without any statistical modelling or adjustment for covariates.
Time Frame: At 1 month post-RSVPreF3 OA vaccine dose administration (at Day 31 for Co-Ad Group and Day 61 for Control Group)
Population: Analysis was performed on PPS for RSVPreF3 OA. Only participants included in 1-month post vaccination timepoint and with data available for RSV-A titers at the specified timepoint were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 388 | 365
Titers | 8119.1 [7316.6 to 9009.7] | 8407.1 [7611.6 to 9285.8]

5. Secondary Outcome: Mean Geometric Increase (MGI) of RSV-A Neutralizing Titers at 1 Month After RSVPreF3 OA Vaccination
Description: The MGI was defined as the geometric mean of the within participant ratios of the post-vaccination titer over the pre-vaccination titer.
Time Frame: At 1 month post-RSVPreF3 OA vaccine dose administration (at Day 31 for Co-Ad Group and Day 61 for Control Group) compared to pre-vaccination (Day 1 for Co-Ad Group and Day 31 for Control Group)
Population: Analysis was performed on PPS for RSVPreF3 OA. Only participants with data available for RSV-A titers at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 382 | 364
Ratio | 8.31 [7.46 to 9.26] | 10.21 [9.20 to 11.33]

6. Secondary Outcome: RSV-A Neutralizing Titers Expressed as Seroresponse Rate (SRR) at 1 Month After RSVPreF3 OA Vaccination
Description: The SRR was defined as the percentage of participants having a fold increase in neutralizing titers (1 month post-study intervention administration over pre-study intervention administration) greater than or equal to (>=) 4.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 282 | 296
Percentage of participants | 73.8 [69.1 to 78.2] | 81.3 [76.9 to 85.2]

7. Secondary Outcome: Percentage of Participants Having RSV-A Neutralizing Titers Greater or Equal to the Assay Cut-off Value at Pre-vaccination and at 1 Month After RSVPreF3 OA Vaccination
Description: Percentage of participants with RSV-A neutralizing titers >= to the assay cut-off value (i.e. lower limit of quantification [LLOQ]) are presented.
Time Frame: At pre-vaccination (Day 1 for Co-Ad Group and Day 31 for Control Group) and at 1 month post-RSVPreF3 OA vaccine dose administration (Day 31 for Co-Ad Group and Day 61 for Control Group)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 406 | 389
Percentage of participants
  At pre-vaccination | 100 [99.1 to 100] | 100 [99.1 to 100]
  1 month post RSVPreF3 administration: number analyzed (Participants) | 388 | 365
  1 month post RSVPreF3 administration | 100 [99.1 to 100] | 100 [99.0 to 100]

8. Secondary Outcome: RSV-B Neutralizing Titers Expressed as GMT at 1 Month After RSVPreF3 OA Vaccination
Description: Neutralizing titers for RSV-B were measured with neutralizing assay and the results were expressed as GMT. GMT is a descriptive statistic calculated directly from the observed titer values at the 1-month post-vaccination timepoint for all participants in the analysis set, without any statistical modelling or adjustment for covariates.
Time Frame: At 1 month post-RSVPreF3 OA vaccine dose administration (at Day 31 for Co-Ad Group and Day 61 for Control Group)
Population: Analysis was performed on PPS for RSVPreF3 OA. Only participants included in 1-month post vaccination timepoint and with data available for RSV-B titers at the specified timepoint were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 388 | 365
Titers | 7537.1 [6791.4 to 8364.5] | 7588.9 [6896.0 to 8351.5]

9. Secondary Outcome: MGI of RSV-B Neutralizing Titers at 1 Month After RSVPreF3 OA Vaccination
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Analysis was performed on PPS for RSVPreF3 OA. Only participants with data available for RSV-B titers at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 382 | 364
Ratio | 6.79 [6.08 to 7.59] | 8.19 [7.35 to 9.12]

10. Secondary Outcome: RSV-B Neutralizing Titers Expressed as SRR at 1 Month After RSVPreF3 OA Vaccination
Description: The SRR was defined as the percentage of participants having a fold increase in neutralizing titers (1 month post-study intervention administration over pre-study intervention administration) >= 4.
Time Frame: as for outcome 5
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 255 | 275
Percentage of participants | 66.8 [61.8 to 71.5] | 75.5 [70.8 to 79.9]

11. Secondary Outcome: Percentage of Participants Having RSV-B Neutralizing Titers Greater or Equal to Assay Cut-off Value at Pre-vaccination and at 1 Month After RSVPreF3 OA Vaccination
Description: Percentage of participants with RSV-B neutralizing titers >= to the assay cut-off value (i.e. LLOQ) are presented.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 406 | 389
Percentage of participants
  At pre-vaccination | 100 [99.1 to 100] | 100 [99.1 to 100]
  1 month post RSVPreF3 administration: number analyzed (Participants) | 388 | 365
  1 month post RSVPreF3 administration | 100 [99.1 to 100] | 100 [99.0 to 100]

12. Secondary Outcome: SARS-CoV-2 Omicron XBB.1.5 Neutralizing Titers Expressed as GMT at 1 Month After COVID-19 mRNA Vaccination
Description: The SARS-CoV-2 Omicron XBB.1.5 neutralizing titers against the pseudovirus bearing S protein were measured with neutralizing assay and the results were expressed as GMT. GMT is a descriptive statistic calculated directly from the observed titer values at the 1-month post-vaccination timepoint for all participants in the analysis set, without any statistical modelling or adjustment for covariates.
Time Frame: At 1 month post-COVID-19 mRNA vaccine dose administration (Day 31 for both groups)
Population: Analysis was performed on PPS for COVID-19 mRNA. Only participants included in 1-month post vaccination timepoint and with data available for SARS-CoV-2 titers at the specified timepoint were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 386 | 388
Titers | 1030.4 [925.2 to 1147.6] | 1407.3 [1244.5 to 1591.4]

13. Secondary Outcome: MGI of SARS-CoV-2 Omicron XBB.1.5 Neutralizing Titers at 1 Month After COVID-19 mRNA Vaccination
Description: as for outcome 5
Time Frame: At 1 month post-COVID-19 mRNA vaccine dose administration (Day 31 for both groups) compared to pre-vaccination (at Day 1 for both groups)
Population: Analysis was performed on PPS for COVID-19 mRNA. Only participants with data available for SARS-CoV-2 Omicron XBB.1.5 neutralizing titers against the pseudovirus bearing S protein at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 380 | 381
Ratio | 4.25 [3.73 to 4.85] | 5.46 [4.74 to 6.30]

14. Secondary Outcome: Percentage of Participants Having SARS-CoV-2 Omicron XBB.1.5 Neutralizing Titers Greater Than or Equal to Assay Cut-off Value at Pre-vaccination and at 1 Month After COVID-19 mRNA Vaccination
Description: Percentage of participants with SARS-CoV-2 Omicron XBB.1.5 neutralizing titers >= to the assay cut-off value (i.e. LLOQ) are presented.
Time Frame: At pre-vaccination (Day 1 for both groups) and at 1 month post-COVID-19 mRNA vaccine dose administration (Day 31 for both groups)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 386 | 388
Percentage of participants
  At pre-dose administration: number analyzed (Participants) | 385 | 381
  At pre-dose administration | 95.1 [92.5 to 97.0] | 94.3 [91.6 to 96.4]
  1 month after COVID-19 mRNA vaccination | 99.7 [98.6 to 100] | 99.7 [98.6 to 100]

15. Secondary Outcome: Number of Participants Reporting Each Solicited Administration Site Event, for Each Type of Vaccine Administered
Description: The solicited administration site events after vaccination included pain, erythema/redness, and swelling. Any = occurrence of the events regardless of the intensity grade.
Time Frame: Within 4 days (the day of administration and 3 subsequent days) after each type of vaccine (RSVPreF3 OA vaccine administered at Day 1 for Co-Ad Group and at Day 31 for Control Group, COVID-19 mRNA vaccine administered at Day 1 for both groups)
Population: Exposed set included all participants in the enrolled set who received at least 1 study intervention. Only those participants with solicited administration site AEs were included in this analysis. Analysis was reported based on each type of vaccine administered (RSVPreF3 OA vaccine and COVID-19 mRNA vaccine).
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 412 | 411
Participants
  Erythema, within 4 days from COVID-19 mRNA Dosing: number analyzed (Participants) | 411 | 411
  Erythema, within 4 days from COVID-19 mRNA Dosing | 19 | 20
  Erythema, within 4 days from RSVPreF3 OA Dosing: number analyzed (Participants) | 412 | 402
  Erythema, within 4 days from RSVPreF3 OA Dosing | 34 | 26
  Pain, within 4 days from COVID-19 mRNA Dosing: number analyzed (Participants) | 411 | 411
  Pain, within 4 days from COVID-19 mRNA Dosing | 297 | 264
  Pain, within 4 days from RSVPreF3 OA Dosing: number analyzed (Participants) | 412 | 402
  Pain, within 4 days from RSVPreF3 OA Dosing | 302 | 235
  Swelling, within 4 days from COVID-19 mRNA Dosing: number analyzed (Participants) | 411 | 411
  Swelling, within 4 days from COVID-19 mRNA Dosing | 10 | 13
  Swelling, within 4 days from RSVPreF3 OA Dosing: number analyzed (Participants) | 412 | 402
  Swelling, within 4 days from RSVPreF3 OA Dosing | 20 | 9

16. Secondary Outcome: Number of Participants Reporting Each Solicited Systemic Event, for Each Day of Dose Administered
Description: The solicited systemic events after vaccination included arthralgia, fatigue, fever (pyrexia), headache and myalgia. Fever was defined as body temperature equal or greater than 38 degrees Celsius (°C). Any = occurrence of the events regardless of the intensity grade.
Time Frame: Within 4 days (the day of dose administered and 3 subsequent days) after each dose (administered at Day 1 for Co-Ad Group and at Days 1 and 31 for Control Group)
Population: Analysis was performed on the Exposed set. Only those participants with solicited systemic AEs were included in this analysis. Analysis was reported based on the day of study dose administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 412 | 411
Participants
  Arthralgia, within 4 days from dosing at Day 1 | 81 | 47
  Arthralgia, within 4 days from dosing at Day 31: number analyzed (Participants) | 0 | 402
  Arthralgia, within 4 days from dosing at Day 31 |  | 36
  Fatigue, within 4 days from dosing at Day 1 | 166 | 115
  Fatigue, within 4 days from dosing at Day 31: number analyzed (Participants) | 0 | 402
  Fatigue, within 4 days from dosing at Day 31 |  | 95
  Fever, within 4 days from dosing at Day 1 | 26 | 7
  Fever, within 4 days from dosing at Day 31: number analyzed (Participants) | 0 | 402
  Fever, within 4 days from dosing at Day 31 |  | 9
  Headache, within 4 days from dosing at Day 1 | 120 | 98
  Headache, within 4 days from dosing at Day 31: number analyzed (Participants) | 0 | 402
  Headache, within 4 days from dosing at Day 31 |  | 83
  Myalgia, within 4 days from dosing at Day 1 | 170 | 117
  Myalgia, within 4 days from dosing at Day 31: number analyzed (Participants) | 0 | 402
  Myalgia, within 4 days from dosing at Day 31 |  | 91

17. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs), for Each Day of Dose Administered
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study vaccine, which does not necessarily have a causal relationship with study vaccine. An unsolicited AE was an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs must had been communicated by participant/participant's caregiver(s) who had signed the informed consent. Unsolicited AEs included both serious and non-serious AEs. Any = occurrence of the events regardless of the intensity grade or relation to study dose administration.
Time Frame: Within 30 days (the day of vaccination and 29 subsequent days) after each dose (dose administered at Day 1 for Co-Ad Group and at Days 1 and 31 for Control Group)
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 417 | 416
Participants
  Within 30 days after dosing at at Day 1 | 87 | 71
  Within 30 days after dosing at at Day 31: number analyzed (Participants) | 0 | 407
  Within 30 days after dosing at at Day 31 |  | 57

18. Secondary Outcome: Number of Participants Reporting Any Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. Any = occurrence of the events regardless of the intensity grade or relation to study dose administration.
Time Frame: Throughout the study period (from Day 1 up to 6 months after the last dose administration [last dose given at Day 1 for Co-Ad Group and Day 31 for Control Group])
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 417 | 416
Participants | 16 | 14

19. Secondary Outcome: Number of Participants Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: The pIMD was defined as a subset of adverse events of special interest that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Any = occurrence of the events regardless of the intensity grade or relation to study dose administration.
Time Frame: as for outcome 18
Population: Analysis was performed on Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 417 | 416
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected within 4 days post each vaccination. Unsolicited AEs were collected within 30 days post each vaccination. All cause mortality, SAEs and pIMDs were collected throughout the study period (from Day 1 up to 6 months post-last administration [last dose given at Day 1 for Co-ad Group and Day 31 for Control Group]).
Description: Solicited and unsolicited events were reported per participant, after any vaccination, for the assessed timeframe according to occurrence of each event, as pre-specified in Statistical Analysis Plan. All events presented in the All-cause mortality, SAE and Other (not including Serious) AEs are reported for the Exposed set.
Arm/Group | Co-Ad Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/417 | 0/416
Serious Adverse Events (participants affected / at risk) | 16/417 | 14/416
Other Adverse Events (participants affected / at risk) | 365/417 | 337/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=417) | Control Group (N=416)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=417) | Control Group (N=416)
Administration site pain (General disorders) | 336 (368) | 303 (499)
Fatigue (General disorders) | 166 (167) | 154 (211)
Administration site erythema (General disorders) | 41 (42) | 36 (46)
Administration site swelling (General disorders) | 25 (26) | 19 (22)
Pyrexia (General disorders) | 26 (26) | 16 (16)
Feeling hot (General disorders) | 3 (3) | 4 (4)
Malaise (General disorders) | 3 (3) | 2 (2)
Chills (General disorders) | 5 (5) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 2 (2)
Administration site pruritus (General disorders) | 2 (2) | 1 (1)
Discomfort (General disorders) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Application site warmth (General disorders) | 0 (0) | 1 (1)
Facial discomfort (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (2)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Administration site rash (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0)
Vaccination site bruising (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 170 (171) | 158 (210)
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 (84) | 73 (88)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 122 (122) | 137 (188)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 5 (5)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 10 (10)
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT06374394/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT06374394/SAP_001.pdf